CLINICAL TRIAL: NCT01855646
Title: Patient Acuity Score With Improved Patient Handoffs to Prevent Sentinel Events
Brief Title: Improved Patient Handoffs to Prevent Sentinel Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00044212
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2014-04

CONDITIONS: Health Care Quality; Access and Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Structured Sign Out Form

SUMMARY:
The overall aim of this project is to improve the quality of the handoffs between hospitalists on the general medicine service at Durham Regional Hospital with the intent of improving transitions of care. The intervention will be an improved and more structured face to face sign-out process using a standardized admission sign-out sheet, which is not part of the official medical record. Daytime admitting physicians will assign an acuity score to their patients in which the severity of illness will be scored from 1-7, with 7 being the most sick / likely to have rapid response team (RRT) or adverse event. The assignment of this score would be based off of the clinician's judgment in the patient's overall assessment. All patients, age >18 years, admitted to the non-resident hospital medicine general medicine service at DRH will be study eligible. Data analysis will examine aggregate hospitalist perception of sign-out practice before and after intervention, total number of RRTs, unplanned transfers, and rapid responses pre and post intervention, percentage of hospitalist based patients of overall rapid responses pre and post intervention, percentage of hospitalists using acuity scores, and average and mean severity score of patients with rapid responses compared with those admitted. Patients have a risk of loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* patients age >18 years
* admitted to the non-resident hospital medicine general medicine service at Durham Regional Hospital (DRH). (This would include transfers from outside hospital, the Emergency Room, intensive care units, and the Durham Rehab Institute.)
* Additionally, hospital medicine faculty who round on the non-resident general medicine service at DRH will be included for the purposes of completion of perception surveys.

Exclusion Criteria:

* Patients presenting for consults, rapid responses handled by surgical services and rapid responses as reason for transfer from Durham Rehabilitation Institute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4344 (Actual)
Dates: Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of RRT's and unplanned transfers pre and post intervention matching aggregate numbers month to month | End of Study, Approximately 6 months

SECONDARY OUTCOMES:
Physician attitudes towards sign-out process pre and post intervention | End of Study, Approximately 6 months

OTHER OUTCOMES:
Compliance rate monthly with sign-out sheet completion; will use simple descriptive statistics | End of Study, Approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Durham Regional Hospital, Durham, North Carolina, United States